CLINICAL TRIAL: NCT06270368
Title: Children Born Preterm: Sustainable Health Monitoring
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Vieri Lastrucci, MD, Meyer Children's Hospital IRCCS
Other Study IDs: PREHMO
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children born preterm are recognized to be at higher risk of short and long term complications and a formal follow-up of infants and children born preterm is recommended by international and national scientific societies. However, in Italy as well as in Tuscany, such a follow up is not usually done, and data are not collected in a structured way. The goal of this observational study is to evaluate the association between a large number of early life exposures and health outcomes and access to care during childhood in infants born preterm. The main questions it aims to answer are: • what is the role of prenatal and perinatal factors in influencing health outcomes during childhood in preterm infants? • What is the role of prenatal and perinatal factors in influencing access to care during childhood? Participants will be asked to attend a follow-up visit for the purpose of collecting health data.

ELIGIBILITY:
Inclusion Criteria:

* Children born preterm (gestational age below 37 weeks at birth) in Tuscany Region
* Acquisition of the informed consent

Exclusion Criteria:

* Residing outside Tuscany region

Ages: 20 Months to 66 Months | Sex: All
Age Groups: Child
Study Population: Preterm infants who were born and reside in the Tuscany region.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant development | The measurements will be assessed at 20-28 months of age
  Infant development comprises physical, cognitive, social-emotional, linguistic, and behavioral milestones. Infant development is assessed with the Bayley Scales Of Infant and Toddler Development third edition (Bayley - III).
Childhood development | The measurements will be assessed at 56-66 months of age
  Childhood development comprises physical, cognitive, social-emotional, linguistic, and behavioral milestones. Childhood development is assessed with the Ages and Stages Questionnaires (ASQ-3).

SECONDARY OUTCOMES:
Presence of visual or hearing impairement | The measurements will be assessed at 20-28 months of age and at 56-66 months of age
Presence of asthma | The measurements will be assessed at 56-66 months of age
Access to care | The measurements will be assessed at 20-28 months of age and at 56-66 months of age
  Hospitalizations and surgeries occurred in the last 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vieri Lastrucci, MD, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (4):
- Italy (4):
  - Azienda Ospedaliero-Universitaria Careggi (AOUC), Florence
  - Meyer Children's Hospital IRCCS, Florence
  - Azienda Ospedaliero Universitaria Pisana (AOUP), Pisa
  - Azienda Ospedaliero Universitaria Senese (AOUS), Siena